CLINICAL TRIAL: NCT01147198
Title: Effectiveness of a Ready-to-Use-Supplementary-Food for the Treatment of Moderate Childhood Malnutrition
Brief Title: Ready to Use Supplementary Food in Moderate Childhood Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medecins Sans Frontieres, Netherlands (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Nutriset (Industry); United Nations World Food Programme (WFP) (Other)
Responsible Party: Pascale Delchevalerie, M.Sc, Medecins Sans Frontieres
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSFOCB1
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2007-03

CONDITIONS: Moderate Acute Malnutrition
Keywords: Moderate; Wasting; Malnutrition; Ready to Use Food; Fortified Blended Flour
MeSH Terms: conditions — Lymphoma, Follicular; Cachexia; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ready to Use Supplementary Food (Active Comparator): Ready to Use Supplementary Food treatment
  Interventions: Dietary Supplement: Ready to Use Supplementary Food
- Premix (Active Comparator): Premix Corn Soy Blend-oil treatment
  Interventions: Dietary Supplement: Premix CSB-oil treatment

INTERVENTIONS:
Dietary Supplement: Ready to Use Supplementary Food — Children received two Supplementary-plumpy® packages per day (184g) providing 1000 Kcal, 26g (10.4%) protein, 68g (61.2%) fat, and 100% of micronutrient requirements based on the Daily Recommended Nutrient Intake.
  Other Names: Supplementary-plumpy®
  Arms: Ready to Use Supplementary Food
Dietary Supplement: Premix CSB-oil treatment — Children received 2 kg of premix per week (226g CSB, 37g oil, and 23g sugar / day) providing 1277 Kcal, 40.7g protein (12.7%), 50.6g (35.7%) fat, and 100% of micronutrient according to the DRNI guidelines
  Other Names: Corn Soy Blend; Fortified Blended Flours
  Arms: Premix

SUMMARY:
Since 2001, Ready to Use Therapeutic Foods (RUTF) are widely used to treat severe malnutrition. Their efficacy and effectiveness were proven in community therapeutic care programs. Recently, the question rose if RUTF would be more effective than enriched flours to treat moderate malnutrition.

The purpose of this study is to compare the effectiveness of Ready to Use Food Supplementary-plumpy® and Premix Corn Soy Blend with oil in term of cure rate, weight gain, duration of treatment, morbidity and mortality in the treatment of moderate acute malnutrition.

Compare the longer term effect on nutritional status and morbidity (relapse?).

ELIGIBILITY:
Inclusion Criteria:

* all children aged 6 months to 5 years admitted to SFC outpatient care during the study period
* WHM between 70-79% (1977 NCHS/WHO standard) without edema
* approval from the caretaker

Exclusion Criteria:

* presence of the following signs: bilateral edema, MUAC<110 mm , WHM< 70%(criteria for severe malnutrition), and medical complications necessitating hospitalisation
* refusal to participate from caretaker

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 570 (Actual)
Dates: Start 2007-04; Primary Completion 2007-08 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Recovery | 112 days
  proportion of children who recovered, defined as WHM> 85% for two consecutive weeks

SECONDARY OUTCOMES:
average weight gain | 112 days
  in g per kg of weight per day
Duration of treatment | 112 days
  average length of stay in days.
Morbidity | 11 months
  number of morbidity episodes during the treatment and six months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Delchevalerie, Msc, Principal Investigator — Medecins Sans Frontieres, Netherlands
Locations (1):
- Health Centers run by MSF and MOH, Bo, Bo, Sierra Leone